CLINICAL TRIAL: NCT05961150
Title: PROMISE: Percutaneous peRipheral cannulatiOn for Minimally-InvaSive Heart Valve surgEry
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PROMISE
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Heart Valve Diseases; Mitral Valve Disease; Aortic Valve Disease; Tricuspid Valve Disease
Keywords: Minimally-invasive heart valve surgery; Percutaneous cannulation; Endovascular closure device
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In addition to conventional heart valve surgery (HVS) via full-sternotomy, which is still the most prevalent therapeutic strategy to address valvular heart disease (VHD), minimally-invasive approaches evolved as safe alternatives, resulting in lower postoperative ventilation times, transfusion rates and shorter in-hospital stay. Femoral artery cannulation is traditionally performed via surgical cutdown to establish cardiopulmonary bypass during minimally-invasive HVS. To avoid groin incision associated infection and lymphocele formation, and further minimize surgical trauma, the use of percutaneous cannulation including novel endovascular closure devices increases as an alternative but remains to be investigated.

The Percutaneous peRipheral cannulatiOn for Minimally-InvaSive heart valve surgEry (PROMISE) registry aims to elucidate the safety, feasibility, and effectiveness of newly developed vascular closure devices during minimally-invasive HVS. Acute intra- and perioperative complications will be evaluated according to modified definitions of the Valve Academic Research Consortium (VARC)-3. In addition, based on the initial results, the comparison of percutaneous cannulation with conventional surgical cut-down techniques is planned.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective analysis of all patients undergoing minimally-invasive heart valve surgery using novel endovascular closure devices for percutaneous cannulation within 6 high-volume heart valve centres in Germany.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Percutaneous peRipheral cannulatiOn for Minimally-InvaSive heart valve surgEry (PROMISE) registry aims to analyse the perioperative outcome of percutaneous peripheral cannulation techniques and their implications during minimally-invasive heart valve surgery.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Access site related vascular complications. | Date of operation (day 0) until 30 days after operation (day 30).
  Incidence (number of) of access site related vascular complications, according to modified Valve Academic Research Consortium 3 (VARC 3) criteria.
All-cause mortality. | Date of operation (day 0) until 30 days after operation (day 30).
  Incidence (number of) of death from any cause.
Cardiovascular mortality. | Date of operation (day 0) until 30 days after operation (day 30).
  Incidence (number of) of cardiovascular death, defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovas-cular accident.

CONTACTS AND LOCATIONS:
Locations (1):
- University Heart and Vascular Center Hamburg, University Medical Centre Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No